CLINICAL TRIAL: NCT05020717
Title: A Multicenter Retrospective Survey of Hyperkalemia Clinical Burden on Hemodialysis Facility-level in China
Brief Title: Retrospective Survey of Hyperkalemia in Hemodialysis
Acronym: Visualize-HD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Li Zuo, Head of the Nephrology Department, Peking University People's Hospital
Other Study IDs: 20-20591
Record Dates: First submitted 2021-08-17; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim to describe hyperkalemia clinical burden and investigate the risk factors associated with the burden on HD facility level.

DETAILED DESCRIPTION:
This study is an observational survey study. We estimate 300 hemodialysis (HD) centres will be enrolled in the study. Summarized data on serum potassium (sK) after long interdialytic interval (LIDI), facility practice pattern and patient characteristics which may be related with sK management, and death records information including number of deaths for each centre will be collected. All the data collected and analysed are on HD facility level, not on patient-level. We are aiming to describe hyperkalemia clinical burden and investigate the risk factors associated with the burden on HD facility level. Association between sK management and long-term outcome will also be explored.

ELIGIBILITY:
Inclusion Criteria:

-

For HD centers:

* ≥ 100 patients under MHD within 3 years prior the study initiation
* Willing to participate in the study
* Have routine blood collection after LIDI
* Have death records

For HD patients:

• On chronic HD for ≥ 3 months

Exclusion Criteria:

* Blood test on other days than those after LIDI
* Unable to provide detailed data required by study protocol
* Being unable to comply with study-specified procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HD centers in China
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the risk factors associated with hyperkalemia clinical burden on HD facility level | 3 years
  Examine the association of risk factors at current status to hyperkalemia prevalence on HD facility level

SECONDARY OUTCOMES:
To describe hyperkalemia clinical burden on HD facility level | 3 years
  Constitution ratio of different sK levels after LIDI in ranges: (0, 3.5], (3.5, 5.0], (5.0, 5.5], (5.5, 6.0], (6.0, 6.5], (6.5, 7.0], (7.0~) mmol/L in HD centers
To describe sK management pattern on HD facility level | 3 years
  Proportion of patients on 3 times/week, 5 times/2 weeks, 2 times/week, less than 2 times/week, and other frequencies of HD treatment Proportion of patients with dialysate potassium concentration at 2.0 mmol/L, 2.5 mmol/L, 3.0 mmol/L and others Proportion of patients with sK testing on monthly, once per 3 months, once per > 3 months and others
To investigate the risk factors associated with crude mortality on HD facility level | 3 years
  Examine the association of risk factors back to 3 years ago to crude mortality on HD facility level, risk factors back to 3 years ago including:
  Constitution ratio of different sK levels after LIDI in ranges: (0, 3.5], (3.5, 5.0], (5.0, 5.5], (5.5, 6.0], (6.0, 6.5], (6.5, 7.0], (7.0~) mmol/L in HD centers back to 3 years ago.
  Constitution ratio of last sK levels before death in ranges: (0, 3.5], (3.5, 5.0], (5.0, 5.5], (5.5, 6.0], (6.0, 6.5], (6.5, 7.0], (7.0~) mmol/L in HD centers Key sK management factors (dialysis frequency, dialysate potassium concentration, sK testing frequency) Other factors (length of dialysis/session, patients dialysis vintage, residual renal function, etiology of ESRD, comorbidities, medication use)

OTHER OUTCOMES:
To investigate the risk factors associated with sK > 6.0 mmol/L and sK > 6.5 mmol/L on HD facility level | 3 years
  Examine the association of the facility-level risk factors at current status with sK ≥ 6.0 mmol/L and ≥ 6.5 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xinju Z, Changying X, Hong L, Guisen L, Ping Z, Caili W, Zuying X, Gang X, Rong W, Rongshan L, Aili J, Hongli J, Jianxin W, Xiaoling W, Jing Y, Li Y, Pei W, Rui Z, Yunhua L, Huimin L, Jinsheng X, Menghua C, Yinhui L, Qinkai C, Zhongfei Y, Yan Z, Hong L, Wenbo H, Chen L, Zhaohui N, Lingling G, Li Z. Prevalence, practice pattern, and mortality of hyperkalemia in Chinese patients undergoing hemodialysis in the visualize HD study. Sci Rep. 2025 Jul 1;15(1):22405. doi: 10.1038/s41598-025-92609-1. PMID 40596462
- [Derived] Zhao X, Zuo L. Multicentre, observational, retrospective cohort of hyperkalaemia burden at haemodialysis facility-level in China: the Visualize-HD study protocol. BMJ Open. 2023 Sep 21;13(9):e066394. doi: 10.1136/bmjopen-2022-066394. PMID 37734899